CLINICAL TRIAL: NCT00034138
Title: A Comparative Pharmacokinetics and Safety Study of OvaRex MAb-B43.13 in Patients With Ovarian Epithelial Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: closed by sponser
Sponsor: Unither Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVA-Gy-16
Record Dates: First submitted 2002-04-23; First posted 2002-04-24 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Ovarian Neoplasms
Keywords: immunotherapy; monoclonal; antibody; Stage III ovarian epithelial cancer; Stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — oregovomab

INTERVENTIONS:
Drug: oregovomab

SUMMARY:
The study will compare the pharmacokinetic profile of OvaRex MAb-B43.13 ascites fluid product and OvaRex MAb-B43.13 cell culture product. Safety and immune responses following treatment with the cell culture product will be evaluated.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, parallel group, Phase 1/2 study in female patients with Stage III/IV epithelial ovarian cancer. The study will compare the pharmacokinetic profile of OvaRex MAb-B43.13 ascites fluid product and OvaRex MAb-B43.13 cell culture product. The study will also evaluate the safety of the cell culture product and the immune responses in patients following treatment. The study is being conducted in three phases:

1. The pharmacokinetic assessment phase will include at least 24 patients, who will be randomized into two treatment groups to receive a single 2 mg dose of either ascites fluid product or cell culture product.
2. The treatment phase will continue administration of two more monthly doses (weeks 4 and 8) and all patients will receive cell culture product. Study patients will be followed for safety and immune response through week 20.
3. The continuation phase will continue administration of cell culture product at the discretion of the investigator on a quarterly schedule for up to 104 weeks in eligible patients who tolerate therapy. Patients who continue treatment will be followed for serious adverse events and all patients will be followed for survival for up to 2 years after first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of epithelial adenocarcinoma of ovarian, tubal or peritoneal origin.
* FIGO Stage III or IV prior to study.
* Serum CA125 level >35 U/mL prior to or at initial surgery. Alternatively, serum CA125 level > or = 100 U/mL following surgery or immunohistochemical evidence of tumor tissue expressing CA125.
* Completed primary treatment following initial diagnosis, including chemotherapy involving a cisplatin or carboplatin-based regimen.
* Functional Performance Status < or = 2 by ECOG scale.
* Medical assessment consistent with prognosis for an expected survival of at least 3 months.
* Voluntary participation, signed informed consent and willingness to complete all study procedures.

Exclusion Criteria:

* No surgery (not including minor surgical procedures), chemotherapy, or radiotherapy (whole abdomen, abdominopelvic or pelvic) within 4 weeks prior to first dose of study drug.
* No known refractory or recurrent disease requiring chemotherapy during the 4 weeks prior to, or planned 10 weeks after first study dose.
* Serum CA125 levels not >800 U/mL at baseline evaluation.
* No gross (clinically evident) ascites.
* No immunotherapy (interferons, tumor necrosis factor, other cytokines or biological response modifiers, or BCG vaccines) within the previous 4 weeks of first study dose.
* No previous treatment with murine monoclonal antibodies for diagnostic or therapeutic purposes or serum human anti-murine antibodies (HAMA) not above upper limit of normal at baseline evaluation.
* Not on long-term chronic treatment with immunosuppressive drugs such as cyclosporin, ACTH, or corticosteroids.
* Ovarian tumors must be of low malignant potential or with noninvasive disease.
* No concurrent malignancy (except non-melanoma of the skin or in situ carcinoma of cervix), unless curative treatment was received and patient has been disease-free for > or = 5 years.
* No known allergy to murine proteins, or prior documented anaphylactic reaction to any drug, or known hypersensitivity to diphenhydramine or other antihistamines of similar chemical structure.
* No previous splenectomy.
* No active autoimmune disease (e.g., rheumatoid arthritis, SLE, ulcerative colitis, Chrohn's Disease, MS, ankylosing spondylitis).
* No recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; no acquired, hereditary, or congenital immunodeficiencies.
* No uncontrolled diseases or illness other than this cancer.
* No significant cardiovascular abnormalities including uncontrolled hypertension, uncontrolled angina, uncontrolled arrhythmias, or CHF (NYHA Classes II-IV).
* No compromised hematopoietic function defined as a hemoglobin <10.0 g/dL or lymphocyte count <300 mm3 or neutrophil count <1000 mm3 or platelet count <100,000 mm3.
* No hepatic dysfunction defined as a bilirubin above upper limit of normal, LDH, SGOT and SGPT >2 times upper limits of normal, or albumin <3.5 g/dL.
* No renal dysfunction defined as serum creatinine above upper limit of normal.
* No pregnancy or breast-feeding (While pregnancy is unlikely in view of the disease and previous surgery, patients who the investigator considers may be at risk of pregnancy will have a pregnancy [beta-HCG] test and will be using a medically approved contraceptive method.)
* No other investigational drugs within 30 days of enrollment.
* No contraindications present to the use of pressor agents.
* No HIV infection, or recent history of drug abuse, alcoholism, or hepatitis.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-03; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Women's Cancer Research Foundation, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - St. Joseph's Medical Center, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia